CLINICAL TRIAL: NCT02285647
Title: An Open-Label, Randomized, Pivotal, Bioequivalence Study of Oral and Intravenous Rolapitant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-11-5016-C
Record Dates: First submitted 2014-09-25; First posted 2014-11-07 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — rolapitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rolapitant - Oral (Experimental): Investigational Product: Rolapitant Dose: 200 mg (4 x 50mg) Route of Administration: Oral Dosage Form: Capsule Dosing Condition: Fasted (10 hours overnight)
  Interventions: Drug: Rolapitant - Oral
- Rolapitant - IV (Experimental): Investigational Product: Rolapitant Dose: 185 mg Route of Administration: IV (30 minutes) Dosage Form: 2 mg/mL solution Dosing Condition: Fasted (10 hours overnight)
  Interventions: Drug: Rolapitant - IV

INTERVENTIONS:
Drug: Rolapitant - Oral — Oral Treatment A Investigational Product: Rolapitant Dose: 200 mg (4 x 50 mg) Route of Administration: Oral Dosage Form: Capsule Dosing Condition: Fasted (10 hours overnight)
  Other Names: Rolapitant
  Arms: Rolapitant - Oral
Drug: Rolapitant - IV — IV Treatment B Investigational Product: Rolapitant Dose: 185 mg Route of Administration: IV (30 minutes) Dosage Form: 2 mg/mL solution Dosing Condition: Fasted (10 hours overnight)
  Other Names: Rolapitant
  Arms: Rolapitant - IV

SUMMARY:
This is an open-label, randomized, single-dose, single-center, parallel-group bioequivalence study of orally- and IV-administered rolapitant in healthy male and female subjects.

DETAILED DESCRIPTION:
To assess the bioequivalence of a single oral dose of 200 mg rolapitant and a single intravenous dose of 185 mg rolapitant administered as an infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be healthy males or females aged 18 to 55 years (inclusive).
2. Female subjects of childbearing potential must have a negative pregnancy test at the Screening visit and on Day -1.
3. Female subjects of childbearing potential must agree to use an accepted method of birth control (excluding hormonal birth control methods) from 72 hours before admission to the clinical unit until study completion.
4. Subjects must have a BMI from 18.5 to 32.0 kg/m2 (inclusive) and a weight of ≥ 50 kg at the Screening visit.
5. Subjects must be able to provide informed consent after risks and benefits have been explained. Subjects must be capable of understanding, able to sign a written informed consent and willing to comply with the protocol requirements.
6. Subjects must be non-tobacco users (defined as a subject who has not smoked or used nicotine products in the last 90 days before administration of study drug) and have a negative cotinine test for nicotine at the Screening visit and Day -1.
7. Subjects must agree to discontinue intake of alcohol and beverages or food known to interfere with CYP metabolic enzymes such as: grapefruit- and quinine-containing food and beverages (e.g., tonic water, bitter lemon), orange juice, prune juice, pomelos, cranberry, pomegranate, star fruit, Seville oranges (or marmalade made from them), garlic supplements, St. John's Wort or licorice from 72 hours before admission to the clinical unit until completion of the study.
8. Subjects must be in general good health as determined by the Investigator, based on prestudy medical and surgical history, physical examination and clinical laboratory tests.
9. Subjects must have cardiovascular (including 12-lead ECG) function at the Screening visit that has no clinically significant abnormalities as determined by the Investigator.

Exclusion Criteria:

1. Subjects who have participated in another investigational study within 30 days or 5 half-lives of the test drug's biologic activity, whichever is longer, before the time of first study dose.
2. Subjects who have a history of hypersensitivity to rolapitant or any of its excipients or who have participated in a previous rolapitant study within 6 months before the time of first study drug dose administration dose (Day 1).
3. Subjects who have a history of relevant allergies (including asthma, food or drug allergies), as determined by the Investigator.
4. Subjects who have had significant blood loss, or have donated or received 1 or more units (450 mL) of blood within 30 days before the first study dose.
5. Subjects who have received any prescription medications or over-the-counter (OTC) medications or herbal supplements within 14 days before the first study dose. By exception, acetaminophen ≤ 1 g/day is permitted.
6. Subjects who have current or recent (within 1 year of the Screening visit) history of alcohol abuse, illicit drug use, physical dependence or addiction to alcohol or any opioid.
7. Cholecystectomized subjects (since biliary excretion is a predominant mode of excretion with rolapitant).
8. Subjects who have any clinical or psychiatric condition or prior therapy that, in the Investigator's opinion, would make the subject unsuitable for the study or unable to comply with the dosing requirements.
9. Subjects who are unwilling or unable to avoid xanthine- and caffeine-containing drinks (including many soft drinks, energy drinks, coffee and tea) and foods (such as chocolate or coffee flavored) from 72 hours before admission through until the subjects are discharged on Day 39.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
AUC0-t: area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration | 39-69 days

SECONDARY OUTCOMES:
Cmax: observed maximum plasma concentration | 39-69 days

OTHER OUTCOMES:
Tmax: observed time to reach Cmax | 39-69 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vargo, MD, Study Director — Tesaro, Inc.
Locations (1):
- Parexel, Baltimore, Maryland, United States